CLINICAL TRIAL: NCT04978194
Title: Effects of an Intervention on University Students' Mental Health and Learning During COVID-19: a Non-randomized Controlled Study
Brief Title: Effects of an Intervention on University Students' Mental Health and Learning During COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nimes (Other)
Responsible Party: Principal Investigator, elodie charbonnier, Associate Professor, University of Nimes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNimes
Record Dates: First submitted 2021-07-22; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Mental Health Issue; Learning Problem; Student Burnout; Motivation; Young Adults/ Students; University-based Intervention
Keywords: Learning; Mental health; Young adults/ Student; University-based Intervention
MeSH Terms: conditions — Burnout, Psychological; Psychological Well-Being | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: During the first academic semester of the academic year 2021/2022, baseline assessments were carried out using an online questionnaire (made on qualtrics secure software) in three groups (online group, hybrid group, control group): measures of mental health (e.g., academic burnout, anxiety and depression), psychological processes (e.g., intolerance of uncertainty, coping, learned helplessness), learning (e.g., cognitive and metacognitive strategies, motivational strategies and beliefs about learning), situational factors (e.g., levels of concern about their health, the health of their loved ones) and socio-demographic factors (e.g., age, level of education, gender, field of study) These assessments were performed in October 2021 (First Time - T1) and December 2021 (Second time - T2).
  During the first academic semester, a university-based intervention to promote better management of emotions and learning was realised in two Experimental group (online group and hybrid group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online group (Experimental): Online group: online university-based 9-weeks intervention to promote better management of emotions and learning. This intervention included:
  1. 9- video capsules (one per week)
  2. An exchange room on each video on a private discord group
  Interventions: Other: University-based intervention to promote better management of emotions and learning
- Hybrid group (Experimental): Hybrid group: hybrid university-based 9-weeks intervention to promote better management of emotions and learning. This intervention included: 10 lessons of 2 hours including
  1. The viewing of the videos
  2. A time of exchange between students, and with the teacher
  Interventions: Other: University-based intervention to promote better management of emotions and learning
- Control group (No Intervention): Control group: No intervention, only two measurement times of 9 weeks apart. Nothing has changed.

INTERVENTIONS:
Other: University-based intervention to promote better management of emotions and learning — It included 9 video capsules (that take place over 9 weeks), with the following themes: stress information, learning information, emotion and stress regulation strategies, cognitive and metacognitive learning strategies, motivation for learning, physical activity, diet, sleep, and managing worry and uncertainty. It is based on previous online student mental health intervention studies. It presents two innovative aspects: elements and examples specific to the COVID-19 pandemic and the addition of modules focused on learning strategies. The different modules were designed by 5 associate professors, 2 Master students in clinical psychology and 2 undergraduate students in psychology. For the control group, the videos will be posted every week on a You Tube channel and broadcast on a private discord group. For the hybrid group, student will have to attend 10 lessons of 2 hours. These courses include the viewing of videos and a time for discussion between students and the teacher.
  Arms: Hybrid group; Online group

SUMMARY:
Since the beginning of the pandemic, several authors (Lee, 2020; Sahu, 2020; Zhai & Du, 2020) have highlighted the various challenges faced by university students, as well as their negative effects on their mental health. A deterioration in their mental health was observed, particularly during lockdown, with very high levels of anxiety and depressive symptoms (Essadek & Rabeyron, 2020; Husky et al., 2020; Le Vigouroux et al., 2021; Odriozola-González et al., 2020). In addition, COVID-19 has brought about a digital revolution in higher education (Strielkowski, 2020). However, distance learning was not without consequences on student stress (IAU, 2020). The detrimental effects of distance education, in terms of stress and anxiety, could also have important consequences for students' learning and academic success.

Our research proposes to evaluate effects of an intervention focused on stress and learning on mental health and learning strategies. This intervention will be proposed to students from University of Nimes. Its primary objective is to prevent psychological health alterations and to improve students' learning strategies.

Three groups will be constituted: a group that will participate in an online program (online group), a group will participate in a hybrid program, i.e. with online content and face-to-face support (hybrid group) and a group that will not be receiving any interventions (control group). The investigators plan to include between 150 and 200 university students, between 40 and 70 in each group.

The levels of mental health and learning strategies of the two experimental group (online and hybrid group) will be compared to a control group with the realization of pre and post intervention measures. Sociodemographic (e.g., level education) and situational variables (e.g., diagnostic of COVID-19) will be considered in the analyses.

DETAILED DESCRIPTION:
In March 2020, the World Health Organization declared the coronavirus disease 2019 (COVID-19) as a global pandemic. In France, all universities have been closed on 16th March 2020. In September 2020, face-to-face teaching restarted in French universities, but with new constraints (e.g., reducing number of students in classrooms, wearing masks) and significant changes in teachings (e.g., distance and/or hybrid education). In October 2020, several French universities closed down again due to significant contamination among students. Finally, on 30th October 2020, the French government imposed a second lockdown and all universities have been closed. It is only in February 2021 that face-to-face teaching started again in French universities (within the limit of 50% of the universities' capacity and 20% of the teachings).

Since the beginning of the COVID-19, a deterioration in their mental health was observed, particularly during lockdown, with very high levels of anxiety and depressive symptoms (Essadek & Rabeyron, 2020; Husky et al., 2020; Le Vigouroux et al., 2021; Odriozola-González et al., 2020). This may be explained in part by the fact that people who were experiencing high levels of psychological distress prior to the pandemic are the most vulnerable (Druss, 2020; Yao et al., 2020), and before COVID-19, university students were already identified as a vulnerable population (see literature review: Paula et al., 2020). Before COVID-19, a central element of students' psychological distress was their difficulties coping with an accumulation of hassles, such as university pressure, schedule changes or financial difficulties (Réveillère et al., 2001). The pandemic confronts students with new and unprecedented events (e.g., online learning, online examinations, regular and significant changes to their schedule) that challenge their ability to adapt (Araújo et al., 2020; Zhai & Du, 2020). Recent research has shown that the more university students used avoidance strategies during lockdown, the more they had symptoms of anxiety and depression (Dawson & Golijani-Moghaddam, 2020; Le Vigouroux et al., 2021). In addition, the inability to tolerate uncertainty in the COVID-19 pandemic can trigger fear of virus (Schimmenti et al., 2020) and impact negatively on psychological well-being (Satici et al., 2020).

COVID-19 has brought about a digital revolution in higher education (Strielkowski, 2020). However, distance learning was not without consequences on student stress (IAU, 2020). This confronts students with new obstacles (e.g., technological, personal, family; Baticulon et al., 2020). The detrimental effects of distance education, in terms of stress and anxiety, could also have important consequences for students' learning and academic success. Indeed, the more depressive and anxiety symptoms learners have, the more their academic difficulties are exacerbated (Mills & Blankstein, 2000), and the less successful their learning strategies are (Warr & Downing, 2000). Furthermore, the fear of losing an academic year was the concern that most exacerbated students' lockdown anxiety (Hasan & Bao, 2020).

The deleterious effects of the pandemic on students' health are now evident. However, some areas of research are still under-explored.

1. Most of the research is largely descriptive and do not identify the factors involved in the deterioration in mental health and learning
2. To date, no interventional studies have been conducted to prevent these deteriorations during the pandemic.

To fill these gaps, our research proposes to evaluate the effects on mental health and learning of a program focused on stress and learning. Our program has been pre-tested during the 2019-2020 academic year. It included nine modules (that take place over 9 weeks) composed of video capsules, with the following themes: stress information, learning information, emotion and stress regulation strategies, cognitive and metacognitive learning strategies, motivation for learning, physical activity, diet, sleep, and managing worry and uncertainty. Particular attention will be paid to the communication tools in order to provide graphic coherence, facilitating the understanding and appropriation of the different media. Our program is based on modules from previous online student mental health intervention studies. It presents, however, two innovative aspects: 1) elements and examples specific to the COVID-19 pandemic and 2) the addition of modules focused on learning strategies. It is therefore an original program, designed within the framework of this research, and adapted to the context of the COVID-19 pandemic (notably concerning the themes of concern, the stressors, or the distance learning courses). The different modules were designed by five associate professors: two specialized in cognitive psychology, experts in learning, two specialized in clinical psychology and cognitive and behavioral therapy, experts in stress and emotion regulation, and one specialized in health psychology, expert in acceptance and commitment therapy. Two Master students in clinical psychology and two undergraduate students in psychology were involved in the process. All the modules are the result of a collaborative effort between the associate professors who contributed their expertise and the students who pre-tested the modules and help improve their design to make them attractive to other students.

For the control group, the videos will be posted every week on a You Tube channel and broadcast on a private discord group. After each video, an associate professor will invite the students to share their feelings, comments, or questions, about the videos in this group. In addition, this researcher will moderate the exchanges. For the hybrid group, student will have to attend 10 lessons of 2 hours. These courses include the viewing of videos and a time for discussion between students and the teacher.

Participants were repeatedly reminded that the program was not a substitute for medical and/or psychotherapeutic care. They were also informed of the services offered by the university (in particular, preventive medicine and health promotion services) which could accompany should they need it. Each participant was identified by a code to aggregate the data between the different measurement times and preserve anonymity. The recruitment was based on voluntary participation and no compensation was offered to participants. The latter signed a consent form and were informed that their information will remain anonymous and their participation was voluntary and could be withdrawn at any time. Measurements are made before and after the intervention, using an online questionnaire (made on qualtrics secure software).

ELIGIBILITY:
Inclusion Criteria:

* Students at the University of Nimes (males and females) aged over 18 years old

Exclusion Criteria:

* not to be a student of the University of Nîmes
* not signing the consent form to participate in the study
* Participants must be in only one group. For example, being in the hybrid group is an exclusion criterion for the online and control group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-25 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety and depressive symptoms | between 5 and 10 minutes
  Units: "mean score". These symptoms are assessed using a French version of the HADS (Lepine et al., 1985). This 14-item self-report questionnaire assesses anxiety symptoms and depressive symptoms (7 items for each dimension) with labels varying from one item to the next. Scores range from 0 to 21 for each dimension, with higher scores reflecting higher levels of anxiety or depressive symptoms. Although this scale has not been specifically validated with students, it is used in many epidemiological studies in the general population to identify the existence of a symptomatology and to assess its severity. This scale presents satisfactory correlations with other scales of depression and anxiety. Internal consistency of the scale is good for anxiety (α between 0.68 and 0.92) and depression (α between 0.67 and 0.90; see the review of Bjelland et al., 2002).
Academic burnout | between 5 and 10 minutes
  Units: "mean score". Academic burnout is measured with the French version of the Maslach Burnout Inventory-General Survey for Students (MBI-GSS; Used with the approval of Mind Garden Inc). This 15-item self-report questionnaire captures 3 dimensions of academic burnout: emotional exhaustion (e.g., "I feel exhausted at the end of a day at the university"), efficacy related to academic work (e.g., "I feel fulfilled when I achieve my academic goals") and cynicism (e.g., "I feel less enthusiastic about my studies"). Each item was assessed using a 7-point Likert-type scale, with responses ranging from 0 (never) to 6 (always). After reverse scoring six items corresponding to the efficacy related to academic work, a high score indicated high academic burnout. Schaufeli et al. (2002) examined the factorial validity and invariance of the MBI-SS with European students and show that the three-factor structure (i.e., exhaustion, cynicism, and efficacy) of the MBI-SS fits to the data.
Cognitive and metacognitive strategies | 5 minutes
  Units: "mean score" and "reported elements". These strategies are measured with visual analog scales ranging from (never) to 100 (all the time) with items asking for the frequency of use in learning practices (e.g., "How well do you plan your study sessions?"), as well as with an open-ended question to assess the methods used by the participant to study in a more qualitative way
Motivational strategies and beliefs | 3 minutes
  Units: "mean score". This dimension is assessed through 8 items related to participants' motivation to learn (2 items; e.g. "How much do you want to start working on your classes?"), their beliefs about learning and intelligence (3 items; e.g. "How much do you consider that making mistakes is a good thing when studying?) and their perceived cognitive load (3 items inspired by Leppink et al. 2013; e.g. "How much do you agree with the following sentence: I will have to concentrate a lot to complete my university studies?). Response labels varied by question but were all in the form of visual analog scales from 0 to 100.

SECONDARY OUTCOMES:
Learned helplessness | between 5 and 10 minutes
  Units: "mean score". Learned helplessness is assessed using a French version of the LHQ which is specific to academic work. Only the subscale measuring learned helplessness was included. Participants rated each of the 12 items on a 5-point Likert scale ranging from Not true to Absolutely true. Higher scores reflected higher levels of an inability to learn. This scale has been validated with Italian students and has good internal reliability (α = .77).
Coping strategies | 10 minutes
  Units: "mean score". Coping are assessed using a French validation of the situational version of the Brief-COPE. Participants were instructed to refer to a stressful situation related to COVID-19 pandemic. This self-report scale assesses fourteen coping strategies (2 items per strategy): active coping, planning, instrumental support, use of emotional support, venting, behavioural disengagement, self-distraction, self-blame, positive reframing, humour, denial, acceptance, religion, and substance use. Participants rated each of the 28 items on a 4-point Likert scale ranging from Never to Always. Higher scores reflected higher levels of strategy use. The French validation of this scale was performed with French students and has good psychometric properties. This scale has good external validity since correlations with instruments assessing psychological balance showed a consistent set of results. It also has good structural validity with the majority of items.
Intolerance of uncertainty | between 5 and 10 minutes
  Units: "mean score". Intolerance of uncertainty is assessed using the French version of the IU Scale - Short Form (Carleton et al., 2007). This self-report scale measures responses to uncertainty, ambiguous situations, and the future. The 12 items are rated on a 5-point Likert scale ranging from 1 ("not at all characteristic of me") to 5 ("entirely characteristic of me"). This scale assesses one total score and two dimensions of the intolerance of uncertainty: the prospective anxiety subscale (with 7 items, e.g., "it frustrates me not having all the information I need"), and inhibitory anxiety subscale (with 5 items, e.g., "when it's time to act, uncertainty paralyses me".) Good convergent and discriminant validity, as well as internal consistency, have been demonstrated by the total score and both subscale scores.
Social support | 5 minutes
  Units: "mean score". Social support is evaluated with the French validation of the Social Provisions Scale-10 item (Caron, 2013). The 10 items are rated on a 4-point Likert scale ranging from 1 ("strongly disagree") to 4 ("Strongly in agreement"). This self-report scale capturing five dimensions of social support (two items per dimension of support): emotional support or attachment (e.g., "I feel a strong emotional bond with at least one other person"), social integration (e.g., "there are people who enjoy the same social activities I do"), reassurance of worth (e.g., "there are people who admire my talents and skills"), tangible help (e.g., "there are people I can count on to help me when I really need it"), and orientation (e.g., "there is someone with whom I can discuss important decisions about my life"). This scale has good psychometric qualities, it is a reliable and valid instrument for measuring the availability of social support.
Well-being | between 5 and 10 minutes
  Units: "mean score". Well-being is evaluated with the French validation (Cottraux, 2009) of the psychological Well-Being Scale (Ryff, 1989). The 18 items are rated on a 6-point Likert scale ranging from 1 ("Disagreement") to 6 ("Agreement"). This self-report scale capturing 6 components of well-being (3 items per components): autonomy ("I tend to be influenced by others when they have strong opinions", control of the environment (e.g., "often, the demands of daily life bring me down"), personal development ("For me, life is a continuous process of learning, change and personal change and personal growth"), positive relationships (e.g., I have not experienced many warm and trusting relationships with others), giving meaning to life (e.g., I live from day to day and don't really think about the future"), and self-acceptance (e.g., I like most aspects of my personality). This scale and its subscales have good psychometric qualities.
Situational factors | 3 minutes
  Six situational factors were considered::
  1. the extent to which participants felt that lockdown was compromising their future job prospects (scale ranging from 0 to 100)
  2. the extent to which university studies were essential to participants (scale ranging from 0 to 100)
  3. the presence or absence of COVID symptoms (dichotomous answer: Yes or No)
  4. the presence or absence of COVID symptoms in their relatives (dichotomous answer: Yes or No)
  5. participants' level of concern about their health owing to the COVID-19 crisis (scale ranging from 0 to 100)
  6. participants' level of concern about their relatives' health owing to the COVID-19 crisis (scale ranging from 0 to 100).
Socio-demographic factors | 2 minutes
  Four socio-demographic factors were considered:
  1. Age
  2. Gender
  3. Level of education
  4. Field of study

CONTACTS AND LOCATIONS:
Locations (1):
- Charbonnier, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charbonnier E, Tremoliere B, Baussard L, Goncalves A, Lespiau F, Philippe AG, Le Vigouroux S. Effects of an online self-help intervention on university students' mental health during COVID-19: A non-randomized controlled pilot study. Comput Hum Behav Rep. 2022 Mar;5:100175. doi: 10.1016/j.chbr.2022.100175. Epub 2022 Feb 10. PMID 35169655
- [Background] Charbonnier, E., Le Vigouroux, S., & Goncalves, A. (2021). Etudiants en temps de confinement et au-delà. La Presse Médicale Formation. https://doi.org/10.1016/j.lpmfor.2021.06.011
- [Result] Le Vigouroux S, Goncalves A, Charbonnier E. The Psychological Vulnerability of French University Students to the COVID-19 Confinement. Health Educ Behav. 2021 Apr;48(2):123-131. doi: 10.1177/1090198120987128. Epub 2021 Jan 20. PMID 33472453
- [Derived] Charbonnier E, Le Vigouroux S, Puechlong C, Montalescot L, Goncalves A, Baussard L, Gisclard B, Philippe AG, Lespiau F. The Effect of Intervention Approaches of Emotion Regulation and Learning Strategies on Students' Learning and Mental Health. Inquiry. 2023 Jan-Dec;60:469580231159962. doi: 10.1177/00469580231159962. PMID 36998220